CLINICAL TRIAL: NCT01335230
Title: Exploring the Role of Gut-associated TH17 in Microbial Translocation in HIV and HCV/HIV Co-infected Patients
Brief Title: The Study of Gut Associated Lymphocytes in HIV and HCV/HIV Co-infected Patients
Status: Completed | Type: Observational
Sponsor: University of Cincinnati (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mohamed Tarek Shata, Principal Investigator, University of Cincinnati
Other Study IDs: UC 10110905
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: HIV; Hepatitis C, Chronic; HCV Coinfection
Keywords: HIV; HCV; Hepatitis C; HIV and Hepatitis C coinfection; HIV/HCV
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Colon tissues
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 10 HIV mono-infected subjects: 10 subjects infected with HIV only
- 10 HCV mono-infected subjects: 10 subjects infected with HCV only
- 10 HIV/HCV co-infected subjects: 10 subjects infected with both HIV and HCV
- 10 control subjects: 10 subjects without HIV, HCV, or both

SUMMARY:
The purpose of this research study is to explore what role immune cells within the gut (the sigmoid colon) have locally and on the immune system of patients infected with HCV, HIV or HCV/ HIV co-infection.

DETAILED DESCRIPTION:
Objective 1: Characterization of the Gut Associated Lymphocytes (GALT) in HIV, HCV and coinfected patients regarding the role of Th17 and cytokine profiles.

Hypothesis 1a: HIV and HCV/HIV coinfection is associated with changes in Th17 numbers and functions in GALT.

Hypothesis 1b: HIV and HCV/HIV coinfection is associated with changes in cytokine profiles in intestinal mucosa.

Objective 2: Identify the relationship between changes in Gut Associated Lymphocytes (GALT) in HIV, HCV and coinfected patients and markers of microbial translocation.

Hypothesis 2a: Changes in GALT are associated with increase in microbial translocation in HIV, HCV and coinfected patients.

ELIGIBILITY:
Inclusion Criteria:

* are at least age 18, but not older than 70 years old
* have HIV, HCV or both
* do not have HIV, HCV or both, and are having a screening colonoscopy or flexible sigmoidoscopy for abdominal pain or colon cancer screening (control subject)

Exclusion Criteria:

* have a history of inflammatory bowel diseases (IBD) or suspected IBD
* have a history of autoimmune diseases including rheumatoid arthritis
* are taking systemic immunomodulators
* are pregnant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll 40 human subjects including 10 HIV mono-infected, 10 HCV mono-infected, 10 HIV/HCV co-infected patients, and 10 control subjects from the outpatient clinic at the University of Cincinnati College of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Tarek Shata, MD, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Shata MT, Abdel-Hameed EA, Hetta HF, Sherman KE. Immune activation in HIV/HCV-infected patients is associated with low-level expression of liver expressed antimicrobial peptide-2 (LEAP-2). J Clin Pathol. 2013 Nov;66(11):967-75. doi: 10.1136/jclinpath-2013-201581. Epub 2013 Aug 12. PMID 23940131
- [Result] Abdel-Hameed EA, Ji H, Sherman KE, Shata MT. Epigenetic modification of FOXP3 in patients with chronic HIV infection. J Acquir Immune Defic Syndr. 2014 Jan 1;65(1):19-26. doi: 10.1097/QAI.0b013e3182a1bca4. PMID 23846566

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled all the planned subjects (40) as suggested in our proposal within 15 months from University of Cincinnati outpatient clinic
Pre-assignment Details: We excluded patients with a history of inflammatory bowel diseases (IBD) or suspected IBD, autoimmune diseases including rheumatoid arthritis, and any patients on systemic immunomodulators. Pregnant women were also excluded from the study.
Period: Overall Study
Arm/Group | 10 HIV Mono-infected Subjects | 10 HCV Mono-infected Subjects | 10 HIV/HCV Co-infected Subjects | 10 Control Subjects
Started | 10 (subjects) | 10 (subjects) | 10 (subjects) | 10 (subjects)
Completed | 10 (subjects) | 10 (subjects) | 10 (subjects) | 10 (subjects)
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 HIV Mono-infected Subjects | 10 HCV Mono-infected Subjects | 10 HIV/HCV Co-infected Subjects | 10 Control Subjects | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (10.7) | 56.8 (6.5) | 49.1 (6.2) | 56 (6.8) | 51.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3 | 6 | 12
  Male | 10 | 7 | 7 | 4 | 28
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Exploring the Role of Gut-associated Th17 in Microbial Translocation in HIV and HCV/HIV Coinfected Patients.
Description: We measure gene transcription of the colon tissues (relative expression fold changes of gene transcription compared to control). No preselected criteria were used to assess the participants. Data were analyzed and compared among each group. Relative expression levels of LEAP-2 (Liver expressed anti-microbial peptide-2) in the four groups were shown in the table below. Detailed of other genes had been published in Shata MT, et al, J. Clin Pathology 2013, Nov 66(11):967-75. PMID 23940131, and Abdel-Hameed et al, J. Acquir Immune Defic Syndr. 2013 Jul 10 PMID: 23846566
Time Frame: One year
Population: All the samples were analyzed for gene array transcriptions and cytokines profiles
Measure: Mean (Standard Deviation); unit: relative expression levels
Arm/Group | 10 HIV Mono-infected Subjects | 10 HCV Mono-infected Subjects | 10 HIV/HCV Co-infected Subjects | 10 Control Subjects
Number analyzed (Participants) | 10 | 10 | 10 | 10
relative expression levels | 5.8 (0.4) | 5.84 (0.5) | 5.84 (0.5) | 6.9 (0.6)

ADVERSE EVENTS:
Arm/Group | 10 HIV Mono-infected Subjects | 10 HCV Mono-infected Subjects | 10 HIV/HCV Co-infected Subjects | 10 Control Subjects
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
small number of subjects enrolled in the study (10 subjects in each group). It is cross-sectional study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No